CLINICAL TRIAL: NCT04652609
Title: Prevention of Chemotherapy-induced Peripheral Neuropathy With Therapeutic Exercise and Blood Flow Restriction Using PRESIONA Program
Brief Title: Preventing Chemotherapy-induced Peripheral Neuropathy Using PRESIONA Exercise Program
Acronym: PRESIONA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRESIONA20
Record Dates: First submitted 2020-10-20; First posted 2020-12-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasm
Keywords: Breast neoplasm; Breast cancer; Therapeutic exercise; Small Fiber Neuropathy
MeSH Terms: conditions — Breast Neoplasms; Small Fiber Neuropathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRESIONA (Experimental): An adapted therapeutic exercise program using blood flow restriction cuff perfomed during chemotherapy treatment. 24-36 sessions of 1 hour multimodal components: aerobic, strength and fascial release exercises. Frequency will be adapted to the recovery status of each patient.
  Interventions: Other: PRESIONA
- Control group (No Intervention): Patients undergoing usual medical treatment

INTERVENTIONS:
Other: PRESIONA — Aerobic and strength exercise combined with restricction blood flow cuffs during chemotherapy treatment
  Other Names: Experimental group; Therapeutic exercise combined with blood flow restriction
  Arms: PRESIONA

SUMMARY:
The aim of this study is to determinate if therapeutic exercise with blood flow restriction (BFR) during neoadjuvant chemotherapy potentialy neurotoxic could prevent the onset of chemotherapy induced peripheral neuropathy (CIPN) comparing to usual care.

DETAILED DESCRIPTION:
CIPN is a side effect of cancer therapies that nowadays has no solution, so our intention is to carry out a preventive therapy against the onset of CIPN. The nature of the studies that try to prevent is very diverse, but one of the wide tools is therapeutic exercise. In this case we intend to combine therapeutic exercise with BFR to obtain a pre-conditioning effect that protects intraepidermal fibers from exposure to the chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* HER2+ breast cancer diagnosis
* On the waiting list to anticancer medical treatment (taxanes-based neoadjuvant chemotherapy)

Exclusion Criteria:

* Previous diagnosis of cancer
* Pregnant
* Cardiac pathology
* No symptoms or pathology that could be confused with neuropathy or related to diabetes
* No recommendation from oncologist for therapeutic exercise practice

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported CIPN symptoms | Change from Baseline to 12 weeks (after intervention)
  Symptoms across to sensory, motor and automic domains will be measured using the questionnarie the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN twenty-item scale. The total questionnaire has a score from 0 to 100, in which a higher score indicates increased symptom burden.

SECONDARY OUTCOMES:
Breast cancer quality of life | Change from baseline to 12 weeks (after intervention)
  assessed by European Organization for Research and Treatment of Breast Cancer-Specific Quality of Life Questionnaire. The total questionnaire has a score from 0 to 100, in which a higher score indicates increased quality of life.
CIPN severity | Change from Baseline to 12 weeks (after intervention)
  assessed by clinical version of The Total Neuropathy Score. Each item is scored from 0 to 4, with the total score ranging from 0 to 24 points; a higher score indicates greater neuropathy severity.
Quality of sleep | Change from Baseline to 12 weeks (after intervention)
  assessed by Pittsburgh Sleep Quality Index that is a self-rated questionnaire which assesses sleep quality and disturbances. The global score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties.
Mood Assessment | Change from Baseline to 12 weeks (after intervention)
  assessed by Scale for Mood Assessment. The scale tries to assess four moods; anxiety, angerhostility, sadness-depression, and happiness. Itd subscale is scory from 0 to 10, a higher score in the EVEA subscales would indicate that the respondent has a higher level of sad-depressed, anxious, angryhostile, and happy mood, respectively.
Pain in hands and feet | Change from Baseline to 12 weeks (after intervention)
  assessed by visual analogue scale. From 0 to 10, a higher score is a worse subjective pain in hands and feet.
Touch Detection Thresholds | Change from Baseline to 12 weeks (after intervention)
  assessed by Semmes-Weinstein filaments (SWMs)
Handgrip strength test | Change from Baseline to 12 weeks (after intervention)
  assessed by TKK5101 Grp-D dynamometer (Takeya, Tokyo, Japan)
General physical functioning and mobility | Change from Baseline to 12 weeks (after intervention)
  assessed by the 6 minutes walking test. A greater distance (meters) covered over 6 min indicates greater mobility and general functioning.
Body composition | Change from Baseline to 12 weeks (after intervention)
  assesseb by bioimpedance (InBody)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero-Villanueva, PhD, Principal Investigator — Physical Therapy Deparment, Faculty of Health Sciences, University of Granada
Locations (1):
- University of Granada, Granada, Spain

REFERENCES:
- [Derived] Lopez-Garzon M, Cantarero-Villanueva I, Legeren-Alvarez M, Gallart-Aragon T, Postigo-Martin P, Gonzalez-Santos A, Lozano-Lozano M, Martin-Martin L, Ortiz-Comino L, Castro-Martin E, Ariza-Garcia A, Fernandez-Lao C, Arroyo-Morales M, Galiano-Castillo N. Prevention of Chemotherapy-Induced Peripheral Neuropathy With PRESIONA, a Therapeutic Exercise and Blood Flow Restriction Program: A Randomized Controlled Study Protocol. Phys Ther. 2022 Mar 1;102(3):pzab282. doi: 10.1093/ptj/pzab282. PMID 35079838